CLINICAL TRIAL: NCT00217269
Title: A Randomized, Controlled Trial of the Medtronic Endeavor Drug (ABT-578) Eluting Coronary Stent System Versus the Taxus Paclitaxel-Eluting Coronary Stent System in De Novo Native Coronary Artery Lesions
Brief Title: The ENDEAVOR IV Clinical Trial: A Trial of a Coronary Stent System in Coronary Artery Lesions
Acronym: ENDEAVOR IV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IP060
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Coronary Artery Disease
Keywords: Restenosis
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Endeavor Drug Eluting Stent
  Interventions: Device: Coronary Artery Stenting
- 2 (Active Comparator): Taxus Drug Eluting Stent
  Interventions: Device: Coronary Artery Stenting

INTERVENTIONS:
Device: Coronary Artery Stenting — Endeavor Drug eluting stent
  Arms: 1
Device: Coronary Artery Stenting — Taxus Drug Eluting Stent
  Arms: 2

SUMMARY:
The purpose of this study is to assess the equivalence in safety and efficacy of the Endeavor Drug Eluting Coronary Stent System when compared to the Taxus Paclitaxel-Eluting Coronary Stent System for the treatment of single de novo lesions in native coronary arteries with a reference vessel diameter (RVD) of 2.5-3.5 mm.

DETAILED DESCRIPTION:
The ENDEAVOR IV Trial is a prospective, multi-center, randomized, two-arm, single-blind trial that will enroll a total of 1,548 patients at up to 80 sites in the US. The ENDEAVOR IV Trial will assess if the Endeavor stent is equivalent in safety and efficacy to the Taxus stent for the treatment of single de novo lesions in native coronary arteries with a RVD of 2.5-3.5 mm.

ELIGIBILITY:
Inclusion Criteria:

* The patient has clinical evidence of ischemic heart disease, stable or unstable angina, silent ischemia, or a positive functional study.
* The patient is an acceptable candidate for percutaneous transluminal coronary angioplasty (PTCA), stenting, and emergent coronary artery bypass graft (CABG) surgery.
* Female patients of childbearing potential must have a negative pregnancy test within 7 days before the procedure.
* The patient or patient's legal representative has been informed of the nature of the study and agrees to its provisions and has provided written informed consent as approved by the Institutional Review Board/Ethics Committee (IRB/EC) of the respective clinical site.
* The patient agrees to return to the same research facility for all required post-procedure follow-up visits.

Exclusion Criteria:

* A known hypersensitivity or contraindication to aspirin, heparin or bivalirudin, ticlopidine or clopidogrel, cobalt, nickel, chromium, molybdenum, polymer coatings (e.g., Phosphorylcholine or Translute), or a sensitivity to contrast media, which cannot be adequately pre-medicated.
* History of an allergic reaction or significant sensitivity to drugs such as ABT-578, rapamycin, tacrolimus, everolimus, or any other analogue or derivative.
* History of an allergic reaction or significant sensitivity to paclitaxel or drugs in similar class.
* A platelet count < 100,000 cells/mm³ or > 700,000 cells/mm³, or a white blood cell (WBC) count < 3,000 cells/mm³.
* A serum creatinine level > 2.0 mg/dl within seven days prior to index procedure.
* Evidence of an acute MI within 72 hours of the intended index procedure (defined as: QWMI or non-Q wave myocardial infarction (NQWMI) having CK enzymes > 2X the upper laboratory normal with the presence of a CK-MB elevated above the Institution's upper limit of normal).
* Previous PCI of the target vessel within 9 months pre-procedure.
* Planned PCI of any vessel within 30 days post-procedure.
* During the index procedure, the target lesion requires treatment with a device other than PTCA prior to stent placement (including but not limited to, cutting balloon, any atherectomy, any laser, thrombectomy, etc.).
* History of a stroke or transient ischemic attack (TIA) within the prior 6 months.
* Active peptic ulcer or upper gastrointestinal (GI) bleeding within the prior 6 months.
* History of bleeding diathesis or coagulopathy or will refuse blood transfusions.
* Concurrent medical condition with a life expectancy of less than 12 months.
* Any previous or planned treatment of the target vessel with anti-restenotic therapies including, but not limited to brachytherapy.
* Currently participating in an investigational drug or another device study that has not completed the primary endpoint or that clinically interferes with the current study endpoints; or requires coronary angiography, IVUS or other coronary artery imaging procedures.
* Documented left ventricular ejection fraction (LVEF) < 30% at most recent evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1548 (Actual)
Dates: Start 2005-04; Primary Completion 2007-03 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Target vessel failure (TVF) rate | 9 months

SECONDARY OUTCOMES:
Angiographic parameters (in-stent and in-segment) including: percent diameter stenosis (%DS) | 8 months
Late lumen loss (in-segment late lumen loss is a powered secondary endpoint) | 9 months
Late loss index | 9 months
Angiographic binary restenosis (ABR) rate | 9 months
Minimum luminal diameter (MLD) | 9 months
Major adverse cardiac event (MACE) rate | 30 days, 6, 9, and 12 months
Neointimal hyperplastic volume and percent volume obstruction (%VO) as measured by intravascular ultrasound (IVUS) | 8 months
Target site revascularization (TSR) rate and clinically-driven TSR rate | 9 months
Target vessel revascularization (TVR) rate and clinically-driven TVR rate | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Martin B. Leon, M.D., Principal Investigator — Columbia University College of Physicians & Surgeons
Locations (1):
- New York-Presbyterian Hospital/Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Derived] Kirtane AJ, Leon MB, Ball MW, Bajwa HS, Sketch MH Jr, Coleman PS, Stoler RC, Papadakos S, Cutlip DE, Mauri L, Kandzari DE; ENDEAVOR IV Investigators. The "final" 5-year follow-up from the ENDEAVOR IV trial comparing a zotarolimus-eluting stent with a paclitaxel-eluting stent. JACC Cardiovasc Interv. 2013 Apr;6(4):325-33. doi: 10.1016/j.jcin.2012.12.123. Epub 2013 Mar 20. PMID 23523453
- [Derived] Mauri L, Massaro JM, Jiang S, Meredith I, Wijns W, Fajadet J, Kandzari DE, Leon MB, Cutlip DE, Thompson KP. Long-term clinical outcomes with zotarolimus-eluting versus bare-metal coronary stents. JACC Cardiovasc Interv. 2010 Dec;3(12):1240-9. doi: 10.1016/j.jcin.2010.08.021. PMID 21232717
- [Derived] Leon MB, Nikolsky E, Cutlip DE, Mauri L, Liberman H, Wilson H, Patterson J, Moses J, Kandzari DE; ENDEAVOR IV Investigators. Improved late clinical safety with zotarolimus-eluting stents compared with paclitaxel-eluting stents in patients with de novo coronary lesions: 3-year follow-up from the ENDEAVOR IV (Randomized Comparison of Zotarolimus- and Paclitaxel-Eluting Stents in Patients With Coronary Artery Disease) trial. JACC Cardiovasc Interv. 2010 Oct;3(10):1043-50. doi: 10.1016/j.jcin.2010.07.008. PMID 20965463
- [Derived] Leon MB, Mauri L, Popma JJ, Cutlip DE, Nikolsky E, O'Shaughnessy C, Overlie PA, McLaurin BT, Solomon SL, Douglas JS Jr, Ball MW, Caputo RP, Jain A, Tolleson TR, Reen BM 3rd, Kirtane AJ, Fitzgerald PJ, Thompson K, Kandzari DE; ENDEAVOR IV Investigators. A randomized comparison of the Endeavor zotarolimus-eluting stent versus the TAXUS paclitaxel-eluting stent in de novo native coronary lesions 12-month outcomes from the ENDEAVOR IV trial. J Am Coll Cardiol. 2010 Feb 9;55(6):543-54. doi: 10.1016/j.jacc.2009.08.067. PMID 20152559
- [Derived] Remak E, Manson S, Hutton J, Brasseur P, Olivier E, Gershlick A. Cost-effectiveness of the Endeavor stent in de novo native coronary artery lesions updated with contemporary data. EuroIntervention. 2010 Feb;5(7):826-32. doi: 10.4244/eijv5i7a138. PMID 20142198
- [Derived] Leon MB, Kandzari DE, Eisenstein EL, Anstrom KJ, Mauri L, Cutlip DE, Nikolsky E, O'Shaughnessy C, Overlie PA, Kirtane AJ, McLaurin BT, Solomon SL, Douglas JS Jr, Popma JJ; ENDEAVOR IV Investigators. Late safety, efficacy, and cost-effectiveness of a zotarolimus-eluting stent compared with a paclitaxel-eluting stent in patients with de novo coronary lesions: 2-year follow-up from the ENDEAVOR IV trial (Randomized, Controlled Trial of the Medtronic Endeavor Drug [ABT-578] Eluting Coronary Stent System Versus the Taxus Paclitaxel-Eluting Coronary Stent System in De Novo Native Coronary Artery Lesions). JACC Cardiovasc Interv. 2009 Dec;2(12):1208-18. doi: 10.1016/j.jcin.2009.10.008. PMID 20129547
- [Derived] Waseda K, Miyazawa A, Ako J, Hasegawa T, Tsujino I, Sakurai R, Yock PG, Honda Y, Kandzari DE, Leon MB, Fitzgerald PJ; ENDEAVOR IV Trial Investigators. Intravascular ultrasound results from the ENDEAVOR IV trial: randomized comparison between zotarolimus- and paclitaxel-eluting stents in patients with coronary artery disease. JACC Cardiovasc Interv. 2009 Aug;2(8):779-84. doi: 10.1016/j.jcin.2009.05.015. PMID 19695548